CLINICAL TRIAL: NCT04229134
Title: Targeting Barriers to Pain Self-Management in Women Veterans: Refinement and Feasibility of a Novel Peer Support Intervention (Project CONNECT) (CDA 18-005)
Brief Title: Piloting a Novel Peer Support Pain Self-Management Intervention (Project CONNECT)
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX 19-003; CDA 18-005 (Other Grant/Funding Number: VA HSRD)
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Musculoskeletal Pain
Keywords: Chronic pain
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilot Arm: Project CONNECT (Other): 8-week home based reciprocal peer support pain self-management program for chronic musculoskeletal pain
  Interventions: Behavioral: Project CONNECT

INTERVENTIONS:
Behavioral: Project CONNECT — Home based pain self-management intervention using peer reinforcement to promote engagement and skill uptake

SUMMARY:
The proposed study will test the feasibility and acceptability of an 8-week home-based reciprocal peer support pain self-management intervention (CONNECT) for women Veterans with chronic musculoskeletal pain. The use of this format will improve the accessibility of treatment to women Veterans who experience logistical, healthcare delivery and psychosocial barriers to care. To address these barriers women Veterans who enroll in CONNECT will be paired and work together to learn/practice pain coping skills, set meaningful activity goals, and participate in a graduated walking program; they will exchange nightly text messages and engage in a weekly 20 minute phone call to reinforce each other and provide support for pain self-management efforts. This is a single-arm pilot project; all eligible and interested women with chronic musculoskeletal pain will receive CONNECT. The primary outcome will be post-treatment and long-term follow-up retention rates.

DETAILED DESCRIPTION:
Objectives: The primary purpose of this pilot study is to evaluate the feasibility and acceptability of a reciprocal peer support pain self-management intervention (CONNECT) for women Veterans with chronic musculoskeletal pain. The primary hypothesis states that the post-treatment and long-term follow-up retention rates will not be less than 80% which is the lowest rate obtained in a behavioral pain trial and comparable to peer support interventions. Several secondary feasibility and acceptability hypotheses are proposed and include: a) rates of successful dyad connection will be greater than or equal to 80%, b) nightly assessment completion rates will meet or exceed the previously established 85% completion rate, c) reported rates of skill practice will meet or exceed 65% consistent with other behavioral pain trials, d) mean intervention satisfaction and credibility ratings will meet or exceed 80% d) 80% or more of participants will report favorable ratings of their peer. A responder analysis will also be completed to determine the percentage of participants who report clinically meaningful reductions in pain intensity and pain interference (as measured by the Brief Pain Inventory- Short Form) and depressive symptoms (as defined by a reduction of 5 or more points on the Patient Health Questionnaire-8). Additional qualitative objectives will solicit participant opinions of candidate control conditions for a future trial.

Research Design: A non-randomized pilot design will be employed. All eligible and interested participants will participate in a week-long behavioral run-in period. Those who successfully navigate it will receive CONNECT. Repeated assessments of key outcome domains will occur at baseline, and at 10 and 22 weeks after intervention start.

Methodology: Participants will be 45 women Veterans with chronic musculoskeletal pain receiving care at the VA Connecticut Healthcare System and VA Central Western Massachusetts. Interested and eligible Veterans will be verbally consented before participating in a brief telephone based qualitative interview and a 1-week behavioral run-in period designed to mimic demands of the intervention/study. Women who successfully navigate the run-in (estimate n=30) will participate in a telephone orientation with their peer and proceed through the 8-week CONNECT intervention. Together, pairs will learn one new pain coping skill each week, participate in a graduated walking program (using a study provided pedometer), and set meaningful activity goals. They will provide reinforcement and support for these activities via text messages and 1 weekly (15 minute call). Study staff will provide periodic feedback on their progress.

ELIGIBILITY:
Inclusion Criteria:

* Women Veteran receiving care at the VA Connecticut Healthcare System or VA Central Western Massachusetts
* Possession of a cell phone with no limits on utilization and willingness to engage in regular phone/text interactions with a peer partner
* Moderate-Severe musculoskeletal pain
* Pain on at least half of the days of the prior six months
* Primary care provider or mental health provider clearance

Exclusion Criteria:

* Life threatening conditions that could impede participation
* Sensory deficits that would impair participation in telephone calls
* Current or pending surgical interventions
* Presence of any mental health condition that would impair ability to engage in treatment or serve as a suitable peer as defined by:

  * diagnosis
  * screening measures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: Retention | 3 months post baseline
  Post-treatment follow-up retention rates and their 95% confidence intervals. These will be compared to 80%, which is the lowest rate obtained in a behavioral pain trial and comparable to peer support interventions
Feasibility: Long-term Retention | 6 months post-baseline
  Long-term follow-up retention rates and their 95% confidence intervals. These will be compared to 80%, which is the lowest rate obtained in a behavioral pain trial and comparable to peer support interventions

SECONDARY OUTCOMES:
Feasibility: Dyad Connection | 3 months post baseline
  Rates of successful dyad connection will be compared to 80% (comparable to other Reciprocal Peer Support interventions)
Feasibility: Diary Completion Rates | 3 months post baseline
  Nightly assessment completion rates and their 95% confidence intervals will be compared to other Veteran behavioral pain trials demonstrating an 85% completion rate.
Feasibility: Skill Practice Rates | 3 months post baseline
  Skill practice rates and their 95% confidence intervals will also be compared to 65% consistent with rates reported in similar pain trials.
Acceptability: Satisfaction & Credibility | 3 months post baseline
  Mean intervention satisfaction and credibility ratings and their 95% confidence intervals will be compared to 80% which is the standard for behavioral pain trials
Acceptability: Peer Matching | 3 months post baseline
  Favorable experience with peer ratings and their 95% confidence intervals will be compared with 80% which is comparable to other reciprocal peer support interventions
Exploratory: Responder Analysis | 3 months post baseline
  A responder analysis will be completed to determine percent of subjects achieving a clinically meaningful reduction in pain intensity, pain interference and depression. For both the Brief Pain Inventory Pain Intensity and Pain Interference subscales, a 30% reduction is defined as clinically meaningful. For depressive symptoms, a reduction of 5 points on the Patient Health questionnaire-8 is considered clinically meaningful
Exploratory: Long-term Responder Analysis | 6 months post baseline
  A responder analysis will be completed to determine percent of subjects achieving a clinically meaningful reduction in pain intensity, pain interference and depression. For both the Brief Pain Inventory Pain Intensity and Pain Interference subscales, a 30% reduction is defined as clinically meaningful. For depressive symptoms, a reduction of 5 points on the Patient Health questionnaire-8 is considered clinically meaningful

CONTACTS AND LOCATIONS:
Overall Officials: Mary Driscoll, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT04229134/ICF_000.pdf